CLINICAL TRIAL: NCT02904837
Title: Mental Practice Combined With Physical Practice to Improve the Gait Performance of People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pikel 01
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2016-09

CONDITIONS: Parkinson Disease
Keywords: Randomized clinical trial; Parkinson's disease; Mental practice; Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (EG) (Experimental): The Experimental training (ET) consists of 10 sessions with 4 blocks of MP (GMP) intercalated with 4 blocks of gait physical practice (GPP), under single (ST) and dual-task (DT) conditions.
  Interventions: Behavioral: Experimental training
- Control Group (Active Comparator): The Control training (CT) consists of 10 sessions with 4 blocks of MP (nGMP) intercalated with 4 blocks of gait physical practice (GPP), under single (ST) and dual-task (DT) conditions.
  Interventions: Behavioral: Control training

INTERVENTIONS:
Behavioral: Experimental training — Each block of MP consists of 5 mental walking attempts with 10 imagined steps. Participants, seated comfortably, eyes closed, will be asked to imagine themselves walking as of a first-person perspective, without any overt physical movement, in four different conditions: habitual speed, as fast as possible, overcoming obstacles and memorizing a name of a specific medication.
  Each block of PP consists of 5 physical walking attempts, with 10 steps. Participants will be asked to walk in 4 different conditions: habitual speed,as fast as possible, overcoming obstacles and memorizing a name of a specific medication.
  Arms: Experimental Group (EG)
Behavioral: Control training — Each block of MP consists of 5 mental walking attempts with 10 imagined steps. Participants, seated comfortably, eyes closed, will be asked to imagine themselves seated appreciating a beautiful landscape as of a first-person perspective, without any overt physical movement, in four different contexts: in a carriage, in a hot air balloon, in a boat and in a zepelin.
  Each block of PP consists of 5 physical walking attempts, with 10 steps. Participants will be asked to walk in 4 different conditions: habitual speed,as fast as possible, overcoming obstacles and memorizing a name of a specific medication.
  Arms: Control Group

SUMMARY:
Among the impairments associated to Parkinson's disease, gait disturbance is one of which that has the most negative impact on the independence in daily living activities and quality of life of people living with Parkinson's disease. Despite the considerable amount of research, we have no consensus about the most efficient physiotherapeutic approach to improve the gait disturbance. Mental practice is considered an efficient strategy to improve the motor performance in healthy individuals and people with stroke. However, there is scarce evidence about its therapeutic results to improve the gait performance in people living with Parkinson's disease. Thus, the aim of this study is to investigate the effects of gait mental practice associated to physical practice to improve the gait performance in people living with Parkinson's disease.

DETAILED DESCRIPTION:
Background: Among the impairments associated to Parkinson's disease, the gait disturbance is one of which that has the most negative impact on the independence in daily living activities and quality of life of people living with Parkinson's disease. Despite the considerable amount of research, we have no consensus about the most efficient physiotherapeutic approach to improve the gait disturbance. Mental practice is considered an efficient strategy to improve the motor performance in healthy individuals and people with stroke. However, there is scarce evidence about its therapeutic results to improve the gait performance in people living with Parkinson's disease.

Objectives: To investigate the effects of mental gait practice associated with physical practice to improve the gait performance of people living with Parkinson's disease.

Design: Parallel, prospective, double-blind, multicentre randomized clinical trial.

Setting: Brazilian Parkinson Association.

Participants: Twenty-two people living with Parkinson's disease in stages 2-3 of disease evolution according to Hoehn and Yahr Classification.

Interventions: The participants will be randomly allocated in an experimental group and a control group. Both groups will perform 10 individual training sessions, two times per week, for five weeks. The training sessions consist of four blocks of mental practice intercalated with four blocks of physical practice of gait under different conditions. The only difference between the groups will be the content of mental practice blocks: the experimental group will perform mental practice of gait while the control group performs non-gait mental practice.

Randomization: Participants will be randomized by ClinStat software into one of two groups: Experimental Group (EG), which will perform gait mental practice; and Control Group (CG), which will perform the non-gait mental practice.

Statistical analysis: The training effects for each primary and secondary outcome measure will be analyzed for the two training conditions (i.e., control and experimental) at the four assessment time points (i.e., pre-intervention, 7 days post-completion and at 30 and 60-day follow-up) using a mixed-design ANOVA with training as the between-group factor and the assessment time point as the within-group factor. The effect sizes (ES) will be calculated for all comparisons at alpha = 0.05. A Tukey HSD post-hoc test will be used for multiple comparisons and p-values below 5 % will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's disease according to the United Kingdom Brain Bank criteria;
* in stage 2-3 of the disease evolution according to the Hoehn and Yahr;
* treated with levodopa or its synergists;
* capable to walk independently indoors without aid;
* referring 5 years of education or more.

Exclusion Criteria:

* presence of other neurological (excluding PD), orthopedic or cardiopulmonary problems;
* visual and auditory deficiency uncorrected;
* dementia [assessed by Montreal Cognitive Assessment (MoCA), cut-off 26];
* depression [according to the Geriatric Depression Scale (GDS-15), cut-off 6];
* declined imagery capacity [according to the Revised Movement Imagery Questionnaire (MIQ-R) cut-off 10].

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Postural Instability and Gait Difficulty Score | up to 3 months
  Postural Instability and Gait Difficulty Score (PIGD): This recommended rating scale for evaluation of gait alterations in PD is based on 5 Unified Parkinson's Disease Rating Scale (UPDRS) items relevant to gait and postural instability (items 13-15, 29, and 30). The 13-15 items are based on gait performance according to PPD perspective, while 29 and 30 items are based on the motor test. It is a recent rating scale that has been used in PD, evaluated independently, which has adequate clinimetric characteristics.
Six-minute Walk Test | up to 3 months
  The six-minute walk test (6-MWT) is a timed recommended clinically based test in which participants are asked to walk for 6 minutes, in their habitual speed, as much distance as possible. Interruptions for resting are permitted if necessary. The 6-MWT has demonstrated adequate test-retest and interrater reliability and minimal detectable change of 82 meters in PD. It may be a good predictor of the ability to independently walk outside safely.
Dynamic Gait Index | up tp 3 months
  The balance during the eight gait related activities is scored in this test. These include quality of walking speed change, going around and over obstacles and stair walking, as well as the number of steps required for a pivot turn.
30-second dual task gait | up tp 3 months
  It measures the maximal walking distance reached in 30 seconds under single task, i.e., without another concurrent task, and dual task, i.e., with a concurrent cognitive task. The cognitive task consists of speaking as many words as possible, starting with a specific character (F, S or A), presented at the beginning of test.

SECONDARY OUTCOMES:
Trail Making Test | up to 3 months
  This test is constituted with two-timed parts: Part A, which involves a visual-scanning task where the participant is required to draw lines sequentially connecting consecutively numbered circles (1-25) randomly arranged on a page as fast as possible. Part B, which assesses cognitive flexibility, where the participant is asked to connect the same number of circles in an alternating sequence of numbers and letters (1, A, 2, B, etc.).
39-item Parkinson's Disease Questionnaire | up to 3 months
  This scale assesses the health-related quality of life, i.e., the impact of an illness and/or treatment on patients' perception of their status of health and on subjective well-being or satisfaction with life. It evaluates 39 parameters in eight groups of issues (mobility, ADL, emotional well-being, stigma of the disease, back in the next, cognitive, communication and bodily discomfort).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, PhD, Principal Investigator — Department of Physioterapy , Communication Science&Disorders, Occupational Therapy, School of Medicine, University of São Paulo
Locations (1):
- Brazil Parkinson Association, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided